CLINICAL TRIAL: NCT03527420
Title: DNA Methylation and Vascular Function in Obesity: Role of Exercise and Weight Loss
Brief Title: DNA Methylation and Vascular Function
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Abeer M. Mohamed, Postdoctoral Research Associate, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2017-1125; 1K99HL140049-01 (NIH)
Record Dates: First submitted 2018-05-03; First posted 2018-05-17 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Obesity; Vascular Dysfunction
Keywords: Obesity; DNA methylation; Exercise; Weight loss; Bariatric; Macrovascular; Microvascular; Epigenetics; Adipose tissue; Adipocytokines; Inflammation; Cardiovascular
MeSH Terms: conditions — Obesity; Motor Activity; Weight Loss; Inflammation | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercising (Active Comparator): 12 weeks of aerobic exercise training
  Interventions: Other: Exercise training
- Non-exercising (No Intervention): standard of care

INTERVENTIONS:
Other: Exercise training — Twelve weeks of aerobic exercise training
  Arms: Exercising

SUMMARY:
The main objective is to examine DNA hypomethylation as an underlying mechanism for the increased production of inflammatory cytokines and the impaired vascular function in obese individuals and as a potential target for nonpharmacological preventive/therapeutic interventions such as aerobic exercise.

DETAILED DESCRIPTION:
The long-term goal of this study is to identify valid targets and strategies for the prevention and treatment of obesity-related cardiovascular disease. Obesity is characterized by a large accumulation of fat tissues that secrete numerous inflammatory mediators (called adipocytokines), generating a systemic inflammatory state. These adipocytokines induce vascular dysfunction which is the initial step towards developing cardiovascular disease. Obesity is affected by environmental factors such as diet and physical activity. These factors induce epigenetic changes, which are changes that affect gene expression without altering the DNA sequence. One of these epigenetic modifications is the reduction in DNA methylation (referred to as hypomethylation) resulting in subsequent increases in gene expression. Preliminary data of the current study showed that the extracted DNA from fat tissues of obese subjects is hypomethylated compared to non-obese controls. DNA hypomethylation correlated significantly with higher expression of adipocytokines and impaired vasodilation in obese subjects. Therefore, the main hypothesis in this study is that the increase in adipocytokine expression in obese adults is mediated by DNA hypomethylation and that DNA hypomethylation is a promising target to prevent obesity-associated inflammation and vascular dysfunction. The flexible modifiable nature of DNA methylation makes it a perfect target for lifestyle interventions such as physical activity and weight loss. Thus, the investigators propose that aerobic exercise training and weight loss following Bariatric surgery will reverse DNA hypomethylation and improve vascular function in obese subjects. This hypothesis will be tested by (1) Investigating abnormal DNA methylation patterns of adipocytokines in fat tissues from obese adults between the age of 18 and 50 compared to non-obese subjects; (2) Test the effectiveness of 12-week aerobic exercise training on reversing DNA hypomethylation and improving vascular function in obese adults; and (3) Examine the effectiveness of weight loss surgery on DNA methylation and vascular function. The proposed studies will improve the understanding of the epigenetic underpinning of obesity-related vascular dysfunction, identify novel therapeutic targets for improving vascular function in obese adults, and provide an evidence for the positive effects of aerobic exercise training and weight loss on the prevention and treatment of obesity-associated cardiovascular disease. These studies will have a positive impact on improving the prevention and therapeutic management of obesity-related cardiovascular morbidities that affect millions of people worldwide.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 35 kg/m2
* Between ages 18-50 years
* Not pregnant
* Approved for a bariatric surgery

Exclusion Criteria:

* To avoid confounding from other inflammatory conditions individuals with current cancer, heart, kidney or liver disease, gallbladder disease or acute or chronic inflammatory diseases (including rheumatoid arthritis, lupus and other autoimmune diseases and genetic diseases) will be excluded
* Pregnant women will be excluded, as they will not be eligible for bariatric surgery
* Current smokers
* Currently abusing alcohol or drugs

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Gender identity
Enrollment: 80 (Estimated)
Dates: Start 2019-10-11 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
DNA methylation status of adipocytokines in obese individuals | Month 24-30
  DNA methylation of 20 preselected adipocytokines using "Amplicon sequencing-based methylation profiling" will be measured in fat tissue collected from obese individuals who are scheduled for bariatric surgery before and after 12 weeks of aerobic exercise training.

SECONDARY OUTCOMES:
Vascular health biomarkers in obese individuals before and after exercise training | Month 24-30
  Serum or plasma levels (pg/ml) of biomarkers of vascular function such as endothelin-1, cyclic guanosine monophosphate (cGMP), and endothelial cell adhesion molecules (soluble intracellular adhesion molecules, soluble vascular cell adhesion molecules, soluble platelet and endothelial cell adhesion molecules, soluble E-selectin, and soluble P-selectin).
Flow induced dilation | Month 1-20
  Measuring reactivity of brachial artery and isolated arterioles from adipose tissues

CONTACTS AND LOCATIONS:
Overall Officials: Abeer Mohamed, MD, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
All data obtained will be shared with the public openly via publication in the most rigorous, visible and appropriate scientific journals possible. Data will be published as soon as it is reasonable to do so (i.e., sufficient data generated to warrant a suitable paper). Supplemental data for each published paper will be made available in one location on the laboratory webpage of the applicant and her mentor. The applicant and other investigators are open to collaboration with outside groups as well when there is mutual interest in this approach. In accordance to the NIH public access requirement (Section 218), we will submit to the National Library of Medicine's PubMed Central an electronic version of our final peer-reviewed manuscripts upon acceptance for publication to be made public no later than 12 months after the official date of publication. We will make every effort to keep findings of this research project widely available and accessible to the research community.
Supporting Information: SAP, CSR
Time Frame: Month 30-36